CLINICAL TRIAL: NCT00031941
Title: A Multidose Phase I Study of Oral CC5013, a Thalidomide Derivative, in Patients With Refractory Metastatic Cancer
Brief Title: CC-5013 in Treating Patients With Cancer That Has Not Responded to Previous Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 020083; 02-C-0083; CDR0000069241; NCT00029081 (obsolete NCT alias)
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Lymphoma; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; unspecified adult solid tumor, protocol specific; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; small intestine lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide

INTERVENTIONS:
Drug: lenalidomide

SUMMARY:
RATIONALE: CC-5013 may stop the growth of cancer by stopping blood flow to the tumor.

PURPOSE: Phase I trial to study the effectiveness of CC-5013 in treating patients who have solid tumors and/or lymphoma that did not respond to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of CC-5013 in patients with refractory solid tumors and/or lymphoma.
* Characterize the pharmacokinetic profile of this drug in these patients.
* Determine whether any correlations can be made between plasma concentrations of this drug and toxicity or clinical activity or biological activity in these patients.
* Characterize the side effect profile of this drug in these patients.
* Determine the dose-limiting toxicity of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oral CC-5013 on day 1. Within 4-10 days, patients begin second course and receive oral CC-5013 once daily on days 1-21. Subsequent courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of CC-5013 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 2 weeks.

PROJECTED ACCRUAL: A total of 3-51 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed refractory solid tumor and/or lymphoma
* No brain metastases or primary CNS malignancies

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* ALT and AST less than 2.5 times normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No unstable or newly diagnosed angina pectoris
* No myocardial infarction within the past 6 months
* No New York Heart Association class II, III, or IV congestive heart failure

Pulmonary:

* No chronic obstructive lung disease requiring oxygen therapy

Other:

* No uncontrolled seizures
* No concurrent acute critical illness
* No serious untreated infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas, mitomycin, or carboplatin)
* No concurrent cytotoxic chemotherapy

Endocrine therapy:

* At least 4 weeks since prior hormonal therapy
* Concurrent luteinizing hormone-releasing hormone agonist required in patients with prostate cancer unless prior orchiectomy has been performed

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* See Endocrine therapy
* Prior surgery allowed

Other:

* Recovered from prior therapy
* No concurrent anticonvulsants (e.g., phenobarbital, phenytoin, or carbamazepine)
* No concurrent rifampin
* No concurrent grapefruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-04; Primary Completion 2007-09 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Dahut, MD, Study Chair — NCI - Medical Oncology Branch
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland

REFERENCES:
- [Background] Tohnya TM, Hwang K, Lepper ER, Fine HA, Dahut WL, Venitz J, Sparreboom A, Figg WD. Determination of CC-5013, an analogue of thalidomide, in human plasma by liquid chromatography-mass spectrometry. J Chromatogr B Analyt Technol Biomed Life Sci. 2004 Nov 25;811(2):135-41. doi: 10.1016/j.jchromb.2004.08.022. PMID 15522712
- [Result] Dahut WL, Aragon-Ching JB, Woo S, Tohnya TM, Gulley JL, Arlen PM, Wright JJ, Ventiz J, Figg WD. Phase I study of oral lenalidomide in patients with refractory metastatic cancer. J Clin Pharmacol. 2009 Jun;49(6):650-60. doi: 10.1177/0091270009335001. PMID 19451403